CLINICAL TRIAL: NCT06454266
Title: Exploration of the Efficacy and Safety of Orelabrutinib Combined With Rituximab and Methotrexate (ORM Regimen) in the First-line Treatment of Primary Central Nervous System Lymphoma
Brief Title: First-line Treatment of PCNSL With the Combination of Orelabrutinib, Rituximab, and Methotrexate (ORM Regimen)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ningbo103
Record Dates: First submitted 2024-05-05; First posted 2024-06-12 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — orelabrutinib; Rituximab; Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ORM regimen(Orelabrutinib, Rituximab and Methotrexate) (Experimental): The subjects received ORM regimen treatment every 21 days for a total of 6 cycles.
  Interventions: Drug: ORM regimen

INTERVENTIONS:
Drug: ORM regimen — The subjects received ORM regimen treatment every 21 days for a total of 6 cycles. The specific medication is as follows " Obutinib tablets 150mg qd d1-21 (suspended 2 days before MTX use until MTX drops to safe concentration) Rituximab 375mg/m2, d1 Methotrexate 3g/m2, d2
  Other Names: Orelabrutinib, Rituximab and Methotrexate

SUMMARY:
Exploring the efficacy and safety of first-line treatment of primary central nervous system lymphoma with the combination of orelabrutinib, rituximab and methotrexate (ORM regimen).

DETAILED DESCRIPTION:
This is an open, single arm, single center clinical study. Untreated primary central nervous system lymphoma patients sign an informed consent form and meet all inclusion criteria. The subjects received treatment with the ORM regimen every 21 days for a total of 6 cycles.

The main purpose is to evaluate the anti-tumor activity (ORR) of the first-line treatment of primary central nervous system lymphoma with the combination of otinib, rituximab, and methotrexate (ORM regimen).

Secondary purpose:

1. Evaluate the safety and tolerability of first-line treatment of primary central nervous system lymphoma with the combination of otinib, rituximab, and methotrexate (ORM regimen).
2. Other efficacy evaluations of the first-line treatment of primary central nervous system lymphoma with the combination of otinib, rituximab, and methotrexate (ORM regimen) include CR, DOR, DCR, and PFS.
3. Evaluate the peripheral blood and cerebrospinal fluid pharmacokinetic characteristics of obrutinib and methotrexate.

The exploratory purpose is to investigate the relationship between the dynamic changes of cerebrospinal fluid ctDNA before and after treatment and the efficacy and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of primary central nervous system lymphoma (PCNSL) of B cell origin，confirmed by pathology (histology or cytology).
2. The patient voluntarily signs the informed consent form.
3. ECOG≤3 points.
4. According to the judgment of the researcher, the expected survival period is more than 3 months.
5. Have measurable lesions, and brain contrast-enhanced MRI shows solid lesions (>10*10mm) ; for those with only meningeal lesions, cytological examination of cerebrospinal fluid (CSF) is required to confirm lymphoma cells and/or imaging findings and CSF examination was consistent.
6. No previous systemic treatment for lymphoma, except corticosteroids;
7. Bone marrow and organ function meet the following standards (no blood transfusion, no use of G-CSF, no use of drug correction within 14 days before screening):

   ① Bone marrow function: Absolute value of neutrophils ≥1.5×109/L, platelets
   * 80×109/L, hemoglobin ≥80g/L;

     * Liver function: serum total bilirubin ≤1.5×ULN (≤3.0×ULN, if there is liver metastasis ); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5.0 × ULN, if there is liver metastasis); ③ Coagulation function: International normalized ratio (INR) and activated partial thrombin time ≤ 1.5 × ULN ;

       * Renal function: Serum creatinine ≤ 1.5 × ULN or estimated creatinine clearance ≥ 60 mL/min (male: Cr (ml/min) = (140-age) × weight (kg) / 72 × serum creatinine concentration (mg/dl) ); Female: Cr (ml/min) = (140-age) × weight (kg)/85 × serum creatinine concentration (mg/dl)).
8. Female subjects of childbearing age and male subjects with childbearing potential who have no childbearing plans with their partners during the study and within 3 months after discontinuing treatment must take one of the following measures during the entire study and within 3 months of discontinuing treatment. Effective contraception: abstinence, physical contraception (such as ligation, condoms, etc.), and the use of hormonal contraceptives should be started at least 3 months before the first dose of medication. Male subjects are prohibited from donating sperm within 3 months from the start of treatment to the end of treatment. The patient or legal guardian voluntarily signed the informed consent form.
9. Good compliance and willingness to comply with visit schedule, dosing plan, laboratory examinations and other test steps.

Exclusion Criteria:

1. The pathological diagnosis was T-cell lymphoma;
2. Have other tumors that require treatment;
3. Uncontrollable active infection;
4. Have uncontrollable or important cardiovascular diseases, including (but not limited to):

   * Any of the following occurring within 6 months before the first dose Conditions: congestive heart failure (NYHA class III or IV), myocardial infarction, unstable angina, or arrhythmia requiring treatment at screening, left ventricular ejection fraction (LVEF) <50%;

     * Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, indeterminate cardiomyopathy); ③ History of clinically significant QTc phase prolongation, II degree type II atrioventricular conduction resistance lag or III degree atrioventricular block or QTc interval (F method) >470msec (female) or >480msec (male); ④ Atrial fibrillation (EHRA grade ≥ 2b); ⑤ Uncontrollable hypertension, as determined by the researcher were judged not to be suitable to participate in this study.
5. Suffering from active hepatitis B or C infection (hepatitis B: acute hepatitis B, untreated chronic hepatitis B virus infection, chronic hepatitis B carriers with HBV-DNA ≥ the detection limit of each center; hepatitis C: HCVRNA positive) or syphilis . Note: Inactive HBV surface antigen (HBsAg) carriers, subjects with active HBV infection and long-lasting anti-HBV suppression (HBV DNA <detection limit of each center), and subjects who have been cured of HCV can be enrolled.
6. HIV-infected patients;
7. Have ever received an organ transplant or allogeneic stem cell transplant.
8. For female subjects, currently in pregnancy or lactation.
9. Those who have previously or currently have pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, etc., and are judged by the researcher to be unsuitable to participate.
10. There have been autoimmune diseases requiring systemic treatment (i.e., disease-modifying antirheumatic drugs, hormones or immunosuppressants) in the past 2 years, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, etc. Rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome-associated vascular thrombosis, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis or glomerulonephritis. The following situations are allowed: autoimmune hypothyroidism or type I diabetes under stable treatment, hormone replacement therapy (such as thyroxine, insulin, or physiological hormone supplementation due to adrenal or pituitary insufficiency) is not considered systemic therapy and is allowed Join the group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Overall response rate | up to 8 months
  Proportion of CR and PR subjects will be assessed at 8 courses

SECONDARY OUTCOMES:
Progress free survival time | up to36 months
  To measure the duration of response over a follow-up period of 36 months
Overall survival | up to36 months
  OS will be assessed from the first receptor given to death or last follow-up
Adverse events profile | up to 8 months
  Number of participants with adverse events. Freguencies of toxicities based on the NCl Common Terminology Critera for AdverseEvents (CTCAE), version 5.0 will be tabulated.
MRD defined by cerebrospinal fluid ctDNA | up to 8 months
  Dynamic changes of cerebrospinal fluid ctDNA before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoying Chen, Principal Investigator — First Affiliated Hospital of Ningbo University
Locations (1):
- The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No